CLINICAL TRIAL: NCT00614159
Title: Ketamine Compared to Propofol for Pediatric GI Endoscopy
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Xiuli Zhang, MD, Upstate Medical University
Other Study IDs: 5545UMU
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-06

CONDITIONS: Endoscopy
Keywords: Child age 1-10 years having a GI Endoscopy with sedation
MeSH Terms: interventions — Ketamine; Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GI Endoscopy
  Interventions: Drug: Ketamine; Drug: Propofol

INTERVENTIONS:
Drug: Ketamine — Weight based dosage for Peds subjects, used for duration of the endoscopy.
Drug: Propofol — Weight based dosage for Peds subjects, used for duration of the endoscopy.

SUMMARY:
Elective outpatient endoscopy for children can be safely performed under general anesthesia with either propofol (1) or ketamine (2) infusions. Both infusions have an advantage over general anesthesia with volatile agents because they do not require intubation. The goal of both infusions is to have the patient breath spontaneously without reacting to the endoscopy which is a noxious stimulus. Patient movement, stridor and vomiting are can interrupt the procedure and increase overall OR time. Propofol also carries the added risk of causing apnea. This side effect is not commonly seen with Ketamine. Our hypothesis is that Ketamine's profile makes it a superior drug to Propofol for elective outpatient endoscopy because of reduced profound intra-operative interruptions and faster recovery time. We plan a study of pediatric patients ages 1 to 10 years old undergoing elective outpatient endoscopy. The patients will be randomized to receiving either a Ketamine or Propofol infusion, and the intra-operative interruptions will be documented by the anesthesiologist. The Post Anesthetic Care Unit (PACU) time to recovery will be monitored and recorded by a third party.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-10
* Endoscopy with sedation scheduled

Exclusion Criteria:

* A history of chronic respiratory disease
* Upper respiratory infection
* Developmental delays
* Dysrhythmias
* Increased intercranial pressure
* Any sedatives or narcotics up to 6 weeks prior to procedure.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pre-op setting, previously scheduled for GI Endoscopy
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)